CLINICAL TRIAL: NCT06453252
Title: Predictors of Intracranial Atherosclerotic Disease in Posterior Circulation: a Cohort Study
Status: Not yet recruiting | Type: Observational
Sponsor: Sohag University (Other)
Collaborators: Emory University (Other)
Responsible Party: Principal Investigator, Mohamed Ahmed Tarek,MD,MSc, Assistant lecturer of Neurology, Sohag University
Other Study IDs: Soh-Med-24-05-04MD
Record Dates: First submitted 2024-06-05; First posted 2024-06-11 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Stroke, Ischemic; Intracranial Atherosclerosis; Posterior Circulation Brain Infarction
MeSH Terms: conditions — Ischemic Stroke; Intracranial Arteriosclerosis; Brain Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- ICAD group: includes ICAD-related stroke made when a smooth-bordered lesions leading to delayed perfusion on conventional-angiography (without competing stroke etiology) or when irregular-surfaced lesions involving the target vessel during mechanical thrombectomy were unveiled (with or without competing stroke etiology).
  Interventions: Other: we are aiming to develop a Scoring system based on certain variables derived from both groups
- Non-ICAD cases (controls): Non-ICAD cases (controls) includes patients with posterior circulation stroke attributed to stroke etiologies other than ICAD.
  Interventions: Other: we are aiming to develop a Scoring system based on certain variables derived from both groups

INTERVENTIONS:
Other: we are aiming to develop a Scoring system based on certain variables derived from both groups — We are aiming to develop a Scoring system based on certain variables derived from both group

SUMMARY:
Early identification of intracranial atherosclerotic disease (ICAD) may impact the management of patients undergoing mechanical thrombectomy (MT). The aim of the study is to develop and validate a scoring system for pre-thrombectomy diagnosis of ICAD in posterior circulation large vessel/distal medium vessel occlusion strokes (LVOs/DMVOs).

ELIGIBILITY:
Inclusion Criteria:

1. Adult ≥18 years
2. Patient with posterior circulation strokes who underwent mechanical thrombectomy.

Exclusion Criteria:

1. Patients with anterior circulation stroke.
2. Patients with intracranial hemorrhage
3. Patients without baseline radiological data.
4. Extracranial large vessel atherosclerosis related strokes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The cohort is divided into 2 groups;
  1. ICAD-related stroke made when a smooth-bordered lesions leading to delayed perfusion on conventional-angiography (without competing stroke etiology) or when irregular-surfaced lesions involving the target vessel during mechanical thrombectomy were unveiled (with or without competing stroke etiology).
  2. Non-ICAD cases (controls) includes patients with posterior circulation stroke attributed to stroke etiologies other than ICAD.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Post-procedural outcomes included any intracranial hemorrhage, symptomatic ICH (sICH) | June 1st, 2025
  sICH is defined as local or remote parenchymal hemorrhage type 2, subarachnoid hemorrhage, and/or intraventricular hemorrhage, combined with a neurological deterioration of 4 points or more on the NIHSS from baseline or leading to death that the physician judged was causative of the deterioration) per ECASS III criteria

SECONDARY OUTCOMES:
90 day modified Rankin scale (mRS) | June 1st, 2025
  a score of 0 to 4 on the modified Rankin scale (range, 0 to 6, with a score of 0 indicating no disability, 4 moderately severe disability, and 6 death) at 90 days, was changed to a good functional status (a modified Rankin scale score of 0 to 3, with a score of 3 indicating moderate disability)
90 day mortality | June 1st, 2025

CONTACTS AND LOCATIONS:
Locations (2):
- Marcus stroke and neuroscience center, Grady Memorial Hospital, Atlanta, Georgia, United States
- Sohag university hospitals, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided